CLINICAL TRIAL: NCT00532116
Title: Pharmacokinetic Comparison of the 6mg/24hr and 12mg/24hr EMSAM (Selegiline Transdermal System) in Healthy Elderly and Non-Elderly Volunteers
Brief Title: PK Comparison of 6mg and 12mg EMSAM in Elderly vs. Non-Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Somerset Pharmaceuticals (Industry)
Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: S9303-P0601
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2007-09-19 (Estimated); Status verified 2007-09

CONDITIONS: Healthy
Keywords: Healthy; Elderly; Non Elderly; Healthy Volunteers
MeSH Terms: interventions — Selegiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): EMSAM 6mg
  Interventions: Drug: EMSAM (Selegiline Transdermal System) 6mg
- B (Active Comparator): EMSAM (Selegiline Transdermal System) 12mg
  Interventions: Drug: EMSAM (Selegiline Transdermal System) 12mg

INTERVENTIONS:
Drug: EMSAM (Selegiline Transdermal System) 6mg — STS 6mg/24hr
  Arms: A
Drug: EMSAM (Selegiline Transdermal System) 12mg — EMSAm 12mg/24Hr
  Arms: B

SUMMARY:
Evaluate the effect of age on the PK of two different doses of EMSAM.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 to 45years of age (inclusive) and 65 years of age or older.
2. Non-obese as defined by being within 15% of desirable body weight for frame size (Appendix II).
3. In general good health as ascertained by physical examination (PE) including measurement of supine and standing vital signs, medical history, clinical laboratory studies, and 12-lead electrocardiogram (ECG).
4. Females must have a negative serum pregnancy test during screening confirmed by a negative urine pregnancy screen at the baseline visit. Women of childbearing potential must agree to continuously use a medically acceptable method of birth control during the course of the study. Acceptable birth control methods are hormonal contraceptives, intrauterine devices or double barrier method (a combination of condom plus contraceptive foam). Postmenopausal females will be eligible to participate if their last normal menses was at least one (1) year prior to study entry.
5. Able and willing to provide informed consent.
6. Able and willing to follow a modified diet.
7. Able and willing to follow the requirements of the study; willing to wear a patch, no swimming, no excessive exercise, etc.

Exclusion Criteria:

1. Presence of significant acute or chronic medical disorder that might complicate or interfere with MAO inhibitor therapy, such as:

   1. Any cardiovascular or cardiac condition requiring drug treatment. Upon review with Sponsor, subjects with well controlled hypertension or hyperlipidemia will be allowed.
   2. History of symptomatic orthostatic hypotension, or in the investigator's best clinicaljudgment a clinically significant postural decrease in systolic blood pressure at screening or baseline.
   3. Type I diabetes mellitus, or poorly controlled Type II diabetes mellitus.
   4. Malignancy and/or chemotherapy within 1 year prior to screening, other than basal cell carcinoma. Malignancies more than 1 year may not preclude participation and will be reviewed on a case-by-case basis by the Somerset Pharmaceuticals, Inc., medical monitor.
   5. Any skin condition (e.g., eczema, psoriasis, dyshydrosis) that might interfere with application and adherence of the STS.
   6. Known or suspected hypersensitivity to selegiline or other MAO inhibitors.
   7. Any significant immunological, pulmonary, hematologic, endocrine and/or metabolic disease or disorder or severe or acute medical illness, that is, metastatic cancer, brain tumors, decompensated cardiac, hepatic or renal failure.
   8. Neurological disorders including delirium, history of head trauma, movement disorders, dementia, multiple sclerosis, stroke, within the past 6 months preceding the study.
2. Any central nervous system disorder including Alzheimer's disease, Parkinson's disease, epilepsy, or cerebrovascular disease.
3. Any psychiatric disorders (except personality disorders).
4. Any mood disorder including MDD which is current or relapsed over the past three years.
5. ADHD.
6. Any conditions that may cause depression including endocrinopathies other than diabetes, lymphoma, pancreatic cancer.
7. Any other illness or disorder that in the opinion of the Investigator would place the subject at significant risk or any inability to follow the requirements of the study regarding maintaining scheduled visits or patch applications.
8. Use of any medication listed below within five half-lives prior to baseline. A longer period of time may be specifically noted for certain medications as indicated:

   1. All contraindicated medications (see Section 7.1.4.3)
   2. Psychotropic medication, including centrally active anticholinergics, anticonvulsants, antiparkinsonian agents, fluoxetine (5 weeks), MAOIs (2 weeks), antipsychotics (oral - 60 days; intramuscular - 10 weeks), anxiolytics, vasodilators (exception: Viagra is permitted), cerebral enhancers (acetylcholinesterase inhibitors), psychostimulants, lithium carbonate, nootropics, reserpine, methyldopa (within 30 days), ergot preparations.
   3. Sympathomimetic drugs, e.g., amphetamines, methylphenidate, dopamine, epinephrine, norepinephrine, over-the-counter (OTC) and prescription nasal decongestants (with the exception of nasal steroids), oral or inhaled sympathomimetic bronchodilators (e.g., albuterol [Proventil], Serevent) and appetite suppressants.
   4. Any serotonergic drug including sumatriptan succinate (Imitrex), zolmitriptan (Zomig), cyproheptadine (Periactin), methysergide (Sansert) or other agonists or antagonists of serotonin receptors.
   5. Meperidine (Demerol), or other opioids.
   6. R(-)tryptophan, metoclopramide.
   7. St. John's wort / hypericum within two (2) weeks and other herbal supplements
   8. Dietary supplements containing tyramine and/or ephedrine.
9. Presence of an Axis-II disorder that makes it unlikely that the subject will be compliant.
10. Presence or history of bipolar disorder or psychotic disorder.
11. Serious risk of suicide.
12. History of substance abuse, including alcohol abuse as defined by DSM-IV criteria, within the past 12 months.
13. Current use of tobacco products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Dose Proportionality of PK parameters and EMSAM release characteristics. | 33 days

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Honolulu, Hawaii, United States